CLINICAL TRIAL: NCT04678115
Title: A Randomized Cross-Over Clinical Trial Comparing Two Non-Surgical Treatments for Severe Blepharoptosis
Brief Title: Clinical Trial Comparing Two Non-Surgical Treatments for Severe Blepharoptosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Principal Investigator, Kevin Houston, Assistant Professor, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2019P003055; R01EY029437 (NIH)
Record Dates: First submitted 2020-12-14; First posted 2020-12-21 (Actual); Results first posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Blepharoptosis; Ptosis, Eyelid; Myasthenia Gravis; Stroke; Traumatic Brain Injury; Chronic Progressive External Ophthalmoplegia
MeSH Terms: conditions — Blepharoptosis; Myasthenia Gravis; Stroke; Brain Injuries, Traumatic; Ophthalmoplegia, Chronic Progressive External

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- MLP first, KTFS second (Experimental): Participants in this arm will receive the MLP in the first period of the crossover and the KTFS in the second period.
  Interventions: Device: Magnetic Levator Prosthesis (MLP); Device: Kinesiotape Frontalis Sling (KTFS)
- KTFS first, MLP second (Experimental): Participants in this arm will receive the KTFS in the first period of the crossover and the MLP in the second period.
  Interventions: Device: Magnetic Levator Prosthesis (MLP); Device: Kinesiotape Frontalis Sling (KTFS)

INTERVENTIONS:
Device: Magnetic Levator Prosthesis (MLP) — Neodymium magnet embedded in a glasses frame and a polymer embedded (PDMS) micro-magnet array fitted externally to the upper lid with IV 3000 securement film. The IV 3000 is FDA approved for extended wear on the skin.
Device: Kinesiotape Frontalis Sling (KTFS) — Kineso Tape is FDA registered as a 510K exempt class 1 device, typically used by physical and occupational therapist to support muscular healing and movement. It is sometimes used on the face in cases of facial palsy or on the eye lid to support the lid in cases of severe blepharoptosis. In such cases it may be attached near the lid margin above the lashes extending up to the forehead skin overlying the frontalis muscle. Alternatively it may be a very short piece attached only along the lid skin. The tape is easily removed.

SUMMARY:
This clinical trial will evaluate two non-surgical devices designed to improve eye lid opening for patients with severe Blepharoptosis (incomplete opening of the eyelids).

DETAILED DESCRIPTION:
Two non-surgical devices for patients with Blepharoptosis will be evaluated. The Magnetic Levator Prosthesis (MLP), is an external device that makes use of a newer class of permanent magnets (made of alloys of neodymium (Nd), iron (Fe) and boron (B)) to restore eyelid movement. The Kinesiotape Frontalis Sling (KTFS), involves the use of tape to help facilitate levator muscle contraction to open the eyelid. Video recordings of spontaneous and volitional blinks will be used to evaluate the effects of each device on eyelid reanimation.

The clinical trial will employ a crossover design in which participants will try each device at home in counterbalanced order with a washout period between. In each period of the crossover, participants will receive training (during study visits at Massachusetts Eye and Ear) in how to apply the device and will then try the device at home for one week with daily follow up by video calls. At the end of the one-week period of home use there will be a study visit at Massachusetts Eye and Ear when the device will be returned and additional video recordings of eye blinks will be made.

At the end of the crossover period, participants will be asked to complete a questionnaire comparing the two devices and to select their preferred device.

ELIGIBILITY:
Inclusion Criteria:

* Presence of ptosis for at least one eye which occludes the visual axis in the resting position (without frontalis drive, lifting with forehead muscles)
* Moderate cognitive function or better defined as greater than or equal to 18 out of 30 on a pre-screening of the Mini-Mental State Exam (MMSE)

Exclusion Criteria:

* Absence of ptosis which occludes the visual axis
* Presence of a corneal ulcer of any size
* Age less than 5 years
* Severe Cognitive impairment defined as MMSE score less than 18, behaviors consistent with delirium (combinations of disorientation, hallucinations, delusions, and incoherent speech), or lethargy.
* Presence of corneal hypoaesthesia;
* Orbicularis weakness on the side of the ptosis
* Mechanical ptosis, including ptosis due to orbital or lid tumor, cicatricial processes affecting the movements of the upper lid, and enophthalmos.
* Previous ptosis surgery less than 3 months prior to Visit 1.
* Lid position affected by lid or conjunctival scarring.
* History of herpes keratitis.
* Periocular neurotoxin (eg, Botox, Xeomin, Dysport, Myobloc) injections on the side of the ptosis within 3 months prior to Visit 1 and during the study.
* History of hyperthyroidism or thyroid eye disease (ie, exophthalmos, upper eyelid retraction, diplopia secondary to extraocular muscle involvement). Hypothyroidism that is controlled on medication is allowed

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Houston, OD MSc, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Upon written request to Massachusetts Eye and Ear data may be provided

REFERENCES:
- [Background] Houston KE, Tomasi M, Yoon M, Paschalis EI. A Prototype External Magnetic Eyelid Device for Blepharoptosis. Transl Vis Sci Technol. 2014 Dec 17;3(6):9. doi: 10.1167/tvst.3.6.9. eCollection 2014 Oct. PMID 25674358
- [Background] Houston KE, Tomasi M, Amaral C, Finch N, Yoon MK, Lee H, Paschalis EI. The Magnetic Levator Prosthesis for Temporary Management of Severe Blepharoptosis: Initial Safety and Efficacy. Transl Vis Sci Technol. 2018 Jan 19;7(1):7. doi: 10.1167/tvst.7.1.7. eCollection 2018 Jan. PMID 29367892
- [Background] Houston KE, Paschalis EI. Feasibility of Magnetic Levator Prosthesis Frame Customization Using Craniofacial Scans and 3-D Printing. Transl Vis Sci Technol. 2022 Oct 3;11(10):34. doi: 10.1167/tvst.11.10.34. PMID 36269183
- [Background] Kurukuti NM, Nadeau M, Paschalis EI, Houston KE. An Adjustable Magnetic Levator Prosthesis for Customizable Eyelid Re-Animation in Severe Blepharoptosis: Design and Proof-of-Concept. Transl Vis Sci Technol. 2023 Aug 1;12(8):11. doi: 10.1167/tvst.12.8.11. PMID 37566397
- [Background] Tirandazi P, Nadeau M, Woods RL, Paschalis EI, Houston KE. An Adjustable Magnetic Levator Prosthesis for Customizable Eyelid Reanimation in Severe Blepharoptosis II: Randomized Evaluation of Angular Translation. Transl Vis Sci Technol. 2023 Dec 1;12(12):1. doi: 10.1167/tvst.12.12.1. PMID 38038607
- [Background] Cheatham SW, Baker RT, Abdenour TE. Kinesiology Tape: A Descriptive Survey of Healthcare Professionals in the United States. Int J Sports Phys Ther. 2021 Jun 1;16(3):778-796. doi: 10.26603/001c.22136. PMID 34123530
- [Background] Lemp MA. Report of the National Eye Institute/Industry workshop on Clinical Trials in Dry Eyes. CLAO J. 1995 Oct;21(4):221-32. No abstract available. PMID 8565190
- [Result] Houston KE, Pundlik S, Shivshanker P, Bowers AR, LaRosa S, Robinson M, Chodosh J, Brandes L, Lee P, Paschalis EI. A Single-Center Sham and Active-Controlled Double-Blind Randomized Crossover Trial of the Magnetic Levator Prosthesis for Severe Blepharoptosis. Transl Vis Sci Technol. 2025 Feb 3;14(2):15. doi: 10.1167/tvst.14.2.15. PMID 39932468

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data for this study were collected at Massachusetts Eye and Ear, Boston, MA. Subjects were recruited by flyer and by referral from other ophthalmology clinics, or neurology clinics.
Pre-assignment Details: One candidate was ruled as ineligible at a pre-screening visit due to lack of blepharoptosis.
Groups:
- MLP First, KTFS Second: Participants in this arm will receive the MLP in the first period of the crossover and the KTFS in the second period.
  This was a cross-over study in which participants received each the Magnetic Levator Prosthesis (MLP) and the Kinesiotape Frontalis Sling (KTFS) devices in counterbalanced order with a washout period between the two interventions. Additionally, the participants also completed a training period for each device prior to the week of at home use, where participants completed baseline assessments with each respective Device and during the MLP training they also underwent assessment using a Sham MLP device.
  Magnetic Levator Prosthesis (MLP): Neodymium magnet embedded in a glasses frame and a polymer embedded (PDMS) micro-magnet array fitted externally to the upper lid with IV 3000 securement film. The IV 3000 is FDA approved for extended wear on the skin.
  Kinesiotape Frontalis Sling (KTFS): Kineso Tape is FDA registered as a 510K exempt class 1 device, typically used by physical and occupational therapist to support muscular healing and movement. It is sometimes used on the face in cases of facial palsy or on the eye lid to support the lid in cases of severe blepharoptosis. In such cases it may be attached near the lid margin above the lashes extending up to the forehead skin overlying the frontalis muscle. Alternatively it may be a very short piece attached only along the lid skin. The tape is easily removed.
- KTFS First, MLP Second: Participants in this arm will receive the KTFS in the first period of the crossover and the MLP in the second period.
  This was a cross-over study in which participants received each the Magnetic Levator Prosthesis (MLP) and the Kinesiotape Frontalis Sling (KTFS) devices in counterbalanced order with a washout period between the two interventions. Additionally, the participants also completed a training period for each device prior to the week of at home use, where participants completed baseline assessments with each respective Device and during the MLP training they also underwent assessment using a Sham MLP device.
  Magnetic Levator Prosthesis (MLP): Neodymium magnet embedded in a glasses frame and a polymer embedded (PDMS) micro-magnet array fitted externally to the upper lid with IV 3000 securement film. The IV 3000 is FDA approved for extended wear on the skin.
  Kinesiotape Frontalis Sling (KTFS): Kineso Tape is FDA registered as a 510K exempt class 1 device, typically used by physical and occupational therapist to support muscular healing and movement. It is sometimes used on the face in cases of facial palsy or on the eye lid to support the lid in cases of severe blepharoptosis. In such cases it may be attached near the lid margin above the lashes extending up to the forehead skin overlying the frontalis muscle. Alternatively it may be a very short piece attached only along the lid skin. The tape is easily removed.
Period: Overall Study
Arm/Group | MLP First, KTFS Second | KTFS First, MLP Second
Started | 9 | 7
Completed | 8 | 7
Not Completed | 1 | 0
Not completed — Lost to Follow-up | 1 | 0

BASELINE CHARACTERISTICS:
Population: The subject that was lost to follow up did not contribute any data to the analysis. No data was collected at their first study visit and so we felt it was best not to report as part of the baseline demographics.
Groups:
- Participants: Baseline characteristics were calculated for the entire group.
Arm/Group | Participants
Number analyzed (Participants) | 15
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 61 [55 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 15
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15
Baseline Interpalpebral Fissure [Mean (Standard Deviation); unit: millimeters] | 3.89 (2.36)

OUTCOME MEASURES:

1. Primary Outcome: Interpalpebral Fissure (IPF) During Spontaneous Blink
Description: The primary outcome was objective measurement of the IPF midpoint height during maximum closing in five spontaneous blinks, captured with a Nikon mirrorless SLR video recording system (Z7II; Nikon USA, Melville, NY, USA), with a visible light source mounted just above the lens, measured manually with ImageJ (National Institutes of Health, Bethesda, MD, USA). Spontaneous blinks are normally incomplete, a behavior that is dependent upon age, gender, task, and environmental demands. Maximum closing was defined as the three points at the base of the blink. Participants were instructed to look at the camera lens and try to relax and behave normally. Recording was stopped after 1 minute or after five spontaneous blinks, whichever came first. Recording always occurred in the same windowless clinical research room with consistent lighting, temperature, humidity, and air flow. The IPF midpoint height during maximum closing in five spontaneous blinks is averaged and reported below.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: millimeters
Groups:
- Magnetic Levator Prosthesis (MLP): Data from when the participants were wearing the MLP.
- Kinesiotape Frontalis Sling (KTFS): Data from when participants were wearing the KTFS.
- Baseline (Sham): Data from when participants were wearing a sham MLP device. Data acts as a baseline + placebo effect.
Arm/Group | Magnetic Levator Prosthesis (MLP) | Kinesiotape Frontalis Sling (KTFS) | Baseline (Sham)
Number analyzed (Participants) | 15 | 15 | 15
millimeters | 2.4 [1.5 to 3.7] | 4.1 [2.6 to 6.5] | 1.1 [0.7 to 1.8]
Statistical Analysis 1: Comparison: Magnetic Levator Prosthesis (MLP) vs Kinesiotape Frontalis Sling (KTFS); Linear mixed-effects regression was used to determine the effect of treatment condition on the spontaneous blink and resting state open IPF, with participant as random intercept. Covariates of age, gender, blink sequence, and crossover order were investigated alone, and significant (P < 0.05) covariates were included in the final model, from which the estimated marginal means and their 95% confidence interval were reported. Hypothesis: MLP allows a more complete spontaneous blink; Test type: Other — Power Calculation: Sample size was estimated based on the treatment condition (three-level factor) effect size on the spontaneous blink IPF measurements (0.55) after eight participants had completed the crossover using one-way analysis of variance power calculation. This led to a sample size of 12 participants with power of 0.80 and type II error of alpha 0.05. To account for possible attrition, 16 were enrolled, with 15 completing the crossover; p < 0.001, Mixed Models Analysis — a priori threshold for statistical significance was p<0.05

2. Secondary Outcome: Interpalpebral Fissure During Resting Open
Description: Resting open IPF was the median between blink-event IPF, measured automatically by a deep learning model for eyelid landmark detection. the IPF midpoint height during resting open was averaged and reported below.
Time Frame: 2 weeks
Measure: Mean (95% Confidence Interval); unit: millimeters
Groups:
- KTFS: Data from when participants were wearing the KTFS.
Arm/Group | Magnetic Levator Prosthesis (MLP) | KTFS | Baseline (Sham)
Number analyzed (Participants) | 15 | 15 | 15
millimeters | 6.8 [5.2 to 8.4] | 7.0 [5.4 to 8.6] | 3.9 [2.3 to 5.5]
Statistical Analysis 1: Comparison: Magnetic Levator Prosthesis (MLP) vs KTFS vs Baseline (Sham); Hypothesis was that both devices (MLP and KFTS) would open the eye equally well, and that both would be better than sham treatment; Test type: Other; p = 0.001, Mixed Models Analysis

3. Secondary Outcome: Proportion of Non-closure During Volitional Blinks
Description: At the end of recording, participants were instructed to close their eyes completely and open completely three times, representing volitional blink trials. These were evaluated manually with ImageJ. Blinks were classified by a human rater as having complete closure, or not, and then the proportion of non-closure blinks across all subjects was calculated for each condition and reported below.
Time Frame: 2 weeks
Measure: Number; unit: Proportion of Non-closure Blinks
Arm/Group | Magnetic Levator Prosthesis (MLP) | KTFS | Baseline (Sham)
Number analyzed (Participants) | 15 | 15 | 15
Proportion of Non-closure Blinks | 0.067 | 0.356 | 0.022
Statistical Analysis 1: Comparison: Magnetic Levator Prosthesis (MLP) vs KTFS vs Baseline (Sham); A test of proportionality was performed to determine the effect of the three treatments on the probability of the eyelid not fully closing; Test type: Other; p = 0.001, test of proportionality

4. Secondary Outcome: Proportion of Subjects Selecting Each Device
Description: Proportion of subjects selecting either the MLP, the KTFS or neither
Time Frame: 6 weeks
Population: All 15 participants were asked to chose which device they liked better, or no device. They were still masked to which was the novel/experimental treatment.
Measure: Count of Participants; unit: Participants
Groups:
- Preferred Magnetic Levator Prosthesis (MLP): Participants who preferred the MLP over KTFS.
- Preferred Kinesiotape Frontalis Sling (KTFS): Participants who preferred KTFS over MLP
- Preferred Neither Treatment: Participants who reported not liking either device.
Arm/Group | Preferred Magnetic Levator Prosthesis (MLP) | Preferred Kinesiotape Frontalis Sling (KTFS) | Preferred Neither Treatment
Number analyzed (Participants) | 15 | 15 | 15
Participants | 7 | 6 | 2

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Magnetic Levator Prosthesis (MLP) | Kinesiotape Frontalis Sling (KTFS) | Baseline (Sham)
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 3/15 | 0/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Magnetic Levator Prosthesis (MLP) (N=15) | Kinesiotape Frontalis Sling (KTFS) (N=15) | Baseline (Sham) (N=15)
Increase in skin erythema scale >3 points (Eye disorders) | 0 (0) | 2 (2) | 0 (0) — Industry skin erythema rating scale
Increase in conjunctival staining >2 points (Eye disorders) | 0 (0) | 1 (1) | 0 (0) — NEI industry scale for ocular surface staining

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-30): https://cdn.clinicaltrials.gov/large-docs/15/NCT04678115/Prot_SAP_000.pdf